CLINICAL TRIAL: NCT02861040
Title: A Phase I Clinical Trial Evaluating the Combination of Volasertib (BI-6727) With Vincristine Sulfate Liposomal Injections (VSLI) in Adult Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia
Brief Title: Volasertib and Vincristine Sulfate Liposome in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Comprehensive Cancer Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16H06; STU00203179 (CTRP (Clinical Trial Reporting Program)); NU 16H06 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01036 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Adult Acute Lymphoblastic Leukemia; Refractory Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; BI 6727

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (volasertib, vincristine sulfate liposome) (Experimental): Patients receive volasertib IV over 1 hour on day 1 and vincristine sulfate liposome IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression, development of an inter-current illness that prevents further administration of treatment, unacceptable toxicity, patient decides to withdraw or treating investigator determines that the patient should be taken off treatment for any reason.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vincristine Sulfate Liposome; Drug: Volasertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo
Drug: Volasertib — Given IV
  Other Names: BI 6727; BI-6727; Polo-like Kinase 1 Inhibitor BI 6727

SUMMARY:
The main purpose of this investigational research study is to determine how safe and tolerable the study drug volasertib is in combination with liposomal vincristine (Marqibo; an FDA-approved drug) in patients with relapsed/refractory acute lymphoblastic leukemia. While VSLI demonstrated an overall response rate of 35% in Acute Lymphoblastic Leukemia (ALL) patients that had failed to respond to or relapsed after chemotherapy, combining it with other agents may increase clinical benefit.

Volasertib inhibits proteins involved in the cell cycle that are increased in ALL. When volasertib inhibits these proteins ALL cells die. In the laboratory, volasertib has been shown to increase activity of vincristine against ALL cells. Therefore, we think the combination of volasertib and VSLI will be more effective against your leukemia than either drug used alone. This study will try to find out what effects, good and/or bad, this drug combination has on the patient and their cancer, and to find a dose that may be used in future studies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of the combination of volasertib and vincristine sulfate liposomal injection (VSLI) in relapsed/refractory (RR) acute lymphoblastic leukemia (ALL).

SECONDARY OBJECTIVES:

I. To determine the toxicity profile of volasertib and VSLI, rate of complete remission (with or without complete hematologic recovery; complete response [CR]/CR with incomplete hematologic recovery [CRi]), duration of remission (DOR), rate of minimal residual disease (MRD)-negativity, progression free survival (PFS), overall survival (OS), 30-day mortality rate.

TERTIARY OBJECTIVES:

I. To determine if volasertib and polo-like kinase (plk)-inhibition down-regulates the mammalian target of rapamycin (mTOR) pathway.

II. Whether plk and mTOR inhibition correlates with clinical response to treatment. III. to determine if volasertib acts synergistically to potentiate the bioavailability and distribution of VSLI.

OUTLINE: This is a dose-escalation study of volasertib.

Patients receive volasertib intravenously (IV) over 1 hour on day 1 and vincristine sulfate liposome IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression, development of an inter-current illness that prevents further administration of treatment, unacceptable toxicity, patient decides to withdraw or treating investigator determines that the patient should be taken off treatment for any reason.

After completion of study, patients are followed up every 28 days for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of Philadelphia-negative ALL by bone marrow biopsy or aspirate
* Patients must have >= 5% blasts in the bone marrow
* Patients must have refractory disease, disease relapse or progression after at least two prior systemic chemotherapy or immunotherapy regimens

  * Note: Exceptions may be made if a patient is deemed unfit for first-line salvage therapy by the treating physician; such cases should be clearly documented
* Patients with a history of CNS (central nervous system) leukemia are eligible if they are not symptomatic from current CNS involvement; if there is CNS involvement that is known prior to enrollment or identified subsequently, it will be treated accordingly with intrathecal chemotherapy per the treating physician
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have adequate organ function within 14 days prior to registration, as defined below:
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/aspartate aminotransferase (ALT) (serum glutamic pyruvic transaminase [SPGT]) =< 3 x ULN
* Creatinine =< 2 X ULN
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test within 14 days prior to registration on study
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy, or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events (=< grade 1 or patient's baseline) due to agents administered more than 2 weeks earlier are not eligible
* Patients may not be receiving any other investigational agents within 7 days of registration
* Patients may not be receiving any medications that are known to prolong QT interval unless reviewed and approved by the principal investigator (PI)
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to volasertib or VSLI are not eligible
* Subject may not have had hematopoietic stem cell transplant (HSCT) meeting any of the following:

  * Is within 2 months of transplant from cycle 1 day 1 (C1D1)
  * Has clinically significant graft-versus-host disease requiring treatment
  * Has >= grade 2 persistent non-hematological toxicity related to the transplant
  * Donor lymphocyte infusion (DLI) is not permitted < 30 days prior to study registration
* Patients with >= grade 2 sensory or motor neuropathy are not eligible
* Fridericia's corrected QT (QTcF) prolongation > 470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome); the QTcF will be calculated as the mean of the 3 electrocardiograms (ECGs) taken at screening

  * NOTE: The formula used to calculate QTcF can be physician's choice, but it must be used consistently throughout the study
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure (>= class 3)
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would, in the investigator's opinion, limit compliance with study requirements
  * Known human immunodeficiency virus (HIV) infection
  * Known John Cunningham virus (JC) virus infection and/or progressive multifocal leukoencephalopathy (PML)
  * Known clinically active hepatitis A, B, or C infections

    * NOTE: Patients with chronic hepatitis C virus (HCV) or hepatitis B virus (HBV) infection may enroll if other laboratory criteria are met; those with HBV surface antigen positivity may enroll only if maintained on appropriate suppressive antiviral therapy for the duration of enrollment in the trial
  * Second malignancy that requires active treatment
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to day 1 of cycle 2
  Determine the MTD of volasertib and VSLI in RR ALL, the MTD will be defined as the highest dose level at which ≤ 1 Dose-Limiting Toxicity (DLT) occurs in 6 patients and will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
Rate of complete remission (CR/Cri) | After every 2 even number cycles during treatment then every 28 days up to 1 year during follow-up
  Evaluate the rate of complete remission (with or without complete hematologic recovery; CR/CRi). Rates will be based on the number and percentage of patients that achieve a CR/CRi. Response will be assessed by bone marrow biopsy and blood counts.
Duration of Remission (DOR) | Up to 1 year from end of treatment
  DOR will be defined from the time, measured in months, of CR or CRi until disease progression.
Minimal Residual Disease (MRD-negativity) rate | Up to 1 year
  The rate of MRD-negativity will be assessed in bone marrow mononuclear cells by multi-color flow cytometry analysis.
Progression Free Survival (PFS) | Up to 1 year from end of treatment
  PFS will be defined as the time from treatment initiation until disease progression.
Overall Survival (OS) | Up to 1 year from end of treatment
  OS is defined as the time from treatment initiation until death from any cause.
30-day mortality rate | Up to 30 days from the first dose of treatment
  Evaluated as the number of patients deceased within the first 30 days from the first dose of treatment.

OTHER OUTCOMES:
Mammalian target of rapamycin (mTOR) protein expression | On cycle 1 day 1 and then 48 hours after 1st volasertib dose
  mTOR phosphoprotein expression levels before and after treatment with volasertib will be analyzed using blood samples which will determine whether protein levels are down-regulated after volasertib exposure.
mTOR phosphoprotein expression levels and clinical response | On cycle 1 day 1 and then 48 hours after 1st volasertib dose
  Assess statistical correlation of decreased mTOR phosphoprotein expression levels with clinical response to treatment with volasertib and VSLI.
Interaction of Volasertib with VSLI in vivo | At day 1 of cycle 1
  Determine if volasertib acts synergistically to potentiate the bioavailability and distribution of VSLI using blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Shira Dinner, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland